CLINICAL TRIAL: NCT00862732
Title: A Randomised Controlled Trial With Cognitive Behavioural Therapy for Persons With Active Suicidal Ideations
Brief Title: Study to Prevent Negative Thoughts of Life
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute for Research & Development Sri Lanka (Other)
Collaborators: Institute of Psychiatry, London (Other)
Responsible Party: Dr Sudath Samaraweera, Principal Investigator, Institute for Research & Development
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRD/03-08
Record Dates: First submitted 2009-03-16; First posted 2009-03-17 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-03

CONDITIONS: Active Suicidal Ideations
Keywords: active suicidal ideation; cognitive behavioural therapy; Sri Lanka; RCT
MeSH Terms: interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 Cognitive Behavioural Therapy (Active Comparator): Intervention group will receive a series of sessions of cognitive behaviour therapy. Delivery of CBT will be by three therapists; PI and two other Medical Officers. Each session will last for 30- 45 minutes and they will be delivered at the participant's residence (or at an alternative place of participant's choice) at two weeks intervals. They will be followed-up for three months from the cessation of CBT sessions.
  Interventions: Behavioral: Cognitive behavioural therapy
- 2 Treatment as usual (Active Comparator): Will be referred to the MO(MH). They also will be followed-up for an equal length of time period as of the participants in the intervention group.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy — Will receive a series of sessions of cognitive behaviour therapy. Delivery of CBT will be by three therapists; PI and two other Medical Officers. Each session will last for 30- 45 minutes and they will be delivered at the participant's residence (or at an alternative place of participant's choice) at two weeks intervals. They will be followed-up for three months from the cessation of CBT sessions.
  Arms: 1 Cognitive Behavioural Therapy
Other: Treatment as usual — Will be referred to the MO(MH). They also will be followed-up for an equal length of time period as of the participants in the intervention group.
  Arms: 2 Treatment as usual

SUMMARY:
The purpose of the study is to test whether cognitive behaviour therapy (CBT) offered by trained therapists, to people with current active suicidal ideations, is efficacious as a secondary prevention strategy in Sri Lanka, when compared with treatment as usual provided by Medical Officers (Mental Health; MO (MH)) of government hospitals

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 64 years
* Self reported current active suicidal ideations
* Ability to speak and write Sinhala

Exclusion Criteria:

* An acute intent and planning of suicide
* In-patient/out-patient treatment following an attempted suicide during the previous two-year period
* A diagnosis of mental retardation
* A diagnosis of sensory deficit
* A diagnosis of alcohol abuse
* A diagnosis of psychotic illness

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
Presence of active suicidal ideations during the follow-up period | three months after the cessation of intervention

SECONDARY OUTCOMES:
Impulsiveness Suicide attempts and completed suicides Client satisfaction Probability of common mental disorders Adherence to treatment regime Retention in the treatment regime Quality of life | three months after the cessation of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Sudath Samaraweera, MBBS MSc MD, Principal Investigator — Institute for Research & Development Sri Lanka
Locations (1):
- Institute for Research & Development, Battaramulla, Sri Lanka